CLINICAL TRIAL: NCT02648971
Title: A Randomized Controlled Trial to Compare Single Portal Versus Two Portal Knee Arthroscopy Techniques in Patients With Meniscal Injuries and Articular Cartilage Pathology
Brief Title: Controlled Trial to Compare Single Versus Two Portal Knee Arthroscopy Techniques
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00030774
Record Dates: First submitted 2015-12-15; First posted 2016-01-07 (Estimated); Results first posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-11

CONDITIONS: Injuries, Knee
Keywords: knee; arthroscopy; portal; meniscus; cartilage injury
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Portal Knee Arthroscopy (Active Comparator): After randomization for each patient is complete, the website will document the name of the person who logged on to perform the randomization, the date and time of the log in, and the surgical group assignment for each patient. This randomization information will be forwarded to the operating room staff so that they can prepare for each study participant's surgical procedure. Patients in Group 1 will undergo knee arthroscopy using a single portal. The details of the surgical procedure for each study participant will be documented on the IKDC Surgical Documentation Form. Study participants in each group will return for standard post-operative follow-up visits at one week, 30 days, and three months. They will return to the clinic at six months and one year for study visits.
  Interventions: Procedure: Single Portal Knee Arthroscopy
- Two Portal Knee Arthroscopy (Active Comparator): Patients in Group 2 will undergo knee arthroscopy using two portals. The details of the surgical procedure for each study participant will be documented on the IKDC Surgical Documentation Form. Study participants in each group will return for standard post-operative follow-up visits at one week, 30 days, and three months. They will return to the clinic at six months and one year for study visits.
  Interventions: Procedure: Two Portal Knee Arthroscopy

INTERVENTIONS:
Procedure: Single Portal Knee Arthroscopy — Patients in Group 1 will undergo knee arthroscopy using a single portal.
  Arms: Single Portal Knee Arthroscopy
Procedure: Two Portal Knee Arthroscopy — Patients in Group 2 will undergo knee arthroscopy using two portals.
  Arms: Two Portal Knee Arthroscopy

SUMMARY:
This randomized, controlled clinical trial will compare the outcomes of single portal versus two portal techniques in patients who have meniscus or articular cartilage pathology. The study hypothesis is that patients who undergo single portal arthroscopy will have less pain post-operatively, use less pain medication, and have a higher International Knee Documentation Committee (IKDC) score at six months and one year compared to patients who undergo traditional two portal knee arthroscopy.

DETAILED DESCRIPTION:
Background, Rationale and Context

Knee arthroscopy procedures provide a minimally invasive method to assess the status of the knee joint in order to repair injuries of the meniscus and articular cartilage. In the past, two or more small openings in the skin (portals) were required in order to allow the passage of both an arthroscope to provide visualization of the knee joint and the instrument used to complete the surgical repair process. However, recent innovations in arthroscopy instrumentation have resulted in the ability to use one portal for knee arthroscopy procedures with both the arthroscope and the instruments passed into the knee joint through the same portal. Both uniportal and two portal arthroscopic techniques are used currently for knee arthroscopy procedures in the Department of Orthopaedic Surgery at Wake Forest Baptist Health.

Objectives

This randomized, controlled clinical trial will compare the outcomes of single portal versus two portal techniques in patients who have meniscus or articular cartilage pathology. The study hypothesis is that patients who undergo single portal arthroscopy will have less pain post-operatively, use less pain medication, and have a higher International Knee Documentation Committee (IKDC) score at six months and one year compared to patients who undergo traditional two portal knee arthroscopy.

Methods and Measures

Design: A randomized, controlled trial

Setting: Academic Medical Center: single study site at Wake Forest Baptist Health

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 21 and 65 years of age, who agree to comply with the protocol
* Patients undergoing a primary knee arthroscopy procedure for meniscus or articular cartilage pathology

Exclusion Criteria:

* Patients with a history of long term pain medication use and/or chronic pain conditions unrelated to the surgery.
* Subjects with severe renal disease, allergies to pain medication, and subjects that will have adverse drug-drug reactions from prescribed pain medication.
* Patients with previous reconstructive procedures, lateral retinacular release, or microfracture
* Active knee infection or sepsis at the time of surgery
* Meniscal injuries requiring repair
* Ligamentous instability
* Advanced degenerative or inflammatory arthritis
* Known cancer at the time of surgery
* Conditions that might interfere with recovery from knee arthroscopy (i.e. conditions or diseases of the nervous and/or muscular system, vascular disease, uncontrolled diabetes)
* Malignant tumor history or treatment of malignant tumor of the knee
* Lower extremity condition causing abnormal ambulation (e.g. ankle fusion, ankle arthroplasty, previous hip fracture, knee arthrofibrosis)
* Pregnant, breast feeding, or planning on becoming pregnant during the time frame of the study, (if a woman of child-bearing age)
* Emotional or neurological conditions that affect the subject's ability or willingness to participate in the study including mental illness or drug and/or alcohol abuse
* Severely overweight (BMI >40) at study enrollment or surgery
* Currently participating in another research study
* Prisoner or impending imprisonment
* Workers' Compensation claims

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth P. Smith, PhD, Study Director — Wake Forest University Health Sciences; John Hubbard, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Irrgang JJ, Anderson AF, Boland AL, Harner CD, Kurosaka M, Neyret P, Richmond JC, Shelborne KD. Development and validation of the international knee documentation committee subjective knee form. Am J Sports Med. 2001 Sep-Oct;29(5):600-13. doi: 10.1177/03635465010290051301. PMID 11573919
- [Background] van de Graaf VA, Wolterbeek N, Scholtes VA, Mutsaerts EL, Poolman RW. Reliability and Validity of the IKDC, KOOS, and WOMAC for Patients With Meniscal Injuries. Am J Sports Med. 2014 Jun;42(6):1408-16. doi: 10.1177/0363546514524698. Epub 2014 Mar 11. PMID 24618098
- [Background] Cooper DE, Fouts B. Single-portal arthroscopy: report of a new technique. Arthrosc Tech. 2013 Jul 19;2(3):e265-9. doi: 10.1016/j.eats.2013.02.017. eCollection 2013. PMID 24265996
- [Background] Crawford K, Briggs KK, Rodkey WG, Steadman JR. Reliability, validity, and responsiveness of the IKDC score for meniscus injuries of the knee. Arthroscopy. 2007 Aug;23(8):839-44. doi: 10.1016/j.arthro.2007.02.005. PMID 17681205

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Portal Knee Arthroscopy | Two Portal Knee Arthroscopy
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Portal Knee Arthroscopy | Two Portal Knee Arthroscopy | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Customized [Count of Participants; unit: Participants]
  0-20 Years old | 0 | 0 | 0
  21-65 Years old | 18 | 18 | 36
  66 and older | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 8 | 11 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-White | 2 | 5 | 7
  White | 16 | 13 | 29
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36
Education [Count of Participants; unit: Participants]
  Less than College Grad | 12 | 8 | 20
  College Grad | 6 | 10 | 16
Activity Level [Count of Participants; unit: Participants]
  Non-Sporting | 9 | 6 | 15
  Sporting | 9 | 12 | 21
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (6.1) | 32.9 (5.0) | 31.6 (5.6)
obese [Count of Participants; unit: Participants] — Population: One subject from the Single Portal Knee Arthroscopy arm and two subjects from the Two Portal Knee Arthroscopy arm did not provide obesity information, which explains the discrepancy in the overall number of participants analyzed for this measure.
  Participants
    Not Obese: number analyzed (Participants) | 17 | 16 | 33
    Not Obese | 8 | 6 | 14
    Obese: number analyzed (Participants) | 17 | 16 | 33
    Obese | 9 | 10 | 19
Smoking Status [Count of Participants; unit: Participants]
  Yes | 2 | 2 | 4
  No | 9 | 11 | 20
  Quit | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: IKDC (International Knee Documentation Committee) Score
Description: IKDC subjective knee evaluation form scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Portal Knee Arthroscopy | Two Portal Knee Arthroscopy
Number analyzed (Participants) | 18 | 18
units on a scale | 36.6 (13.3) | 40.2 (11.1)

2. Primary Outcome: IKDC Score
Description: as for outcome 1
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Portal Knee Arthroscopy | Two Portal Knee Arthroscopy
Number analyzed (Participants) | 18 | 18
units on a scale | 55.7 (21.6) | 57.5 (19.6)

3. Primary Outcome: IKDC Score
Description: as for outcome 1
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Portal Knee Arthroscopy | Two Portal Knee Arthroscopy
Number analyzed (Participants) | 18 | 18
units on a scale | 63.1 (25.6) | 66.7 (24.0)

4. Primary Outcome: IKDC Score
Description: as for outcome 1
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Portal Knee Arthroscopy | Two Portal Knee Arthroscopy
Number analyzed (Participants) | 18 | 18
units on a scale | 61.5 (23.4) | 67.4 (19.7)

5. Primary Outcome: IKDC Score
Description: as for outcome 1
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Portal Knee Arthroscopy | Two Portal Knee Arthroscopy
Number analyzed (Participants) | 18 | 18
units on a scale | 64.1 (25.6) | 72.6 (12.7)

6. Secondary Outcome: Pain Levels
Description: Pain levels will also be collected at the 1 and 4 day telephone calls. Range 0 - 10, higher scores denotes worse outcomes
Time Frame: Days 1 and 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Portal Knee Arthroscopy | Two Portal Knee Arthroscopy
Number analyzed (Participants) | 18 | 18
units on a scale
  Day 1 | 3.6 (2.2) | 3.9 (2.7)
  Day 4 | 2.0 (1.6) | 2.5 (2.3)

7. Secondary Outcome: Number of Participants That Required the Use of Pain Medication
Time Frame: Days 1 and 4
Measure: Count of Participants; unit: Participants
Arm/Group | Single Portal Knee Arthroscopy | Two Portal Knee Arthroscopy
Number analyzed (Participants) | 18 | 18
Participants
  Day 1 | 15 | 13
  Day 4 | 10 | 6

8. Secondary Outcome: Number of Participants That Required the Use of Narcotics
Time Frame: Days 1 and 4
Measure: Count of Participants; unit: Participants
Arm/Group | Single Portal Knee Arthroscopy | Two Portal Knee Arthroscopy
Number analyzed (Participants) | 18 | 18
Participants
  Day 1 | 13 | 11
  Day 4 | 7 | 4

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Single Portal Knee Arthroscopy | Two Portal Knee Arthroscopy
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT02648971/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT02648971/Prot_SAP_001.pdf